CLINICAL TRIAL: NCT00512876
Title: Effectiveness and Safety of Topical Bevacizumab (Avastin) for Treatment of Corneal Neovascularization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Michael J. Mines, MD, Research Director, Ophthalmology, Walter Reed Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRAMC WU# 07-23022
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Corneal Neovascularization
MeSH Terms: conditions — Corneal Neovascularization | interventions — Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab (Avastin) — Bevacizumab 10mg/mL 1 drop BID x 3 weeks

SUMMARY:
Purpose: To determine the efficacy and safety of one commonly used VEGF inhibitor, bevacizumab (Avastin, Genentech), as a topical agent for the treatment of corneal neovascularization.

ELIGIBILITY:
Inclusion Criteria:

* male or female, at least 18 years of age
* clinically stable corneal neovascularization
* superficial or deep corneal neovascularization that extends farther than 2mm from the limbus
* ability to understand and provide informed consent to participate in this study and willingness to follow study instructions and likely to complete all required visits.

Clinical stability - all of the following criterial should be excluded before a corneal neovascularization can be regarded as clinically stable:

* current or recent (<3 months) episode of corneal and ocular surface infection (bacterial, viral, fungal, or acanthamoebal)
* recent (<3 months) ocular surgery, including cataract surgery, and/or laser of any type in the study eye
* recent (<6 months) full thickness or lamellar keratoplasty
* recent (<6 months) ocular surface reconstruction, limbal auto or allograft stem cell transplantation, or amniotic membrane transplantation
* current or recent (<3 months) use of contact lens or plan to use contact lens (excluding bandage contact lens)
* current or recent (<3 months) persistent corneal epithelial defect (of at leat 14 days duration) measuring more than 1mm2

Exclusion Criteria:

* current or recent (<1 month) systemic corticosteroid therapy or periocular corticosteroid injections to the study eye
* current or recent (<3 months) intravitreal durg injection to the study eye.
* recent (<1 month) change in dose and frequency of topical steroids and/or non-steroidal anti-inflammatory agents
* uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic blood pressure of >90 mmHg
* history of a thromboembolic event, including myocardial infarction or cerebral vascular accident
* patients age 75 or older
* history of renal abnormalities
* recent (<3 months) or planned surgery
* history of coagulation abnormalities, including end stage liver disease or current anticoagulation medication other than aspirin (warfarin, heparin, enoxaparin or similar anticoagulant agent)
* all female patients of childbearing potential will be excluded. A female is considered to be of childbearing potential unless she is postmenopausal and without menses for 12 months or without a uterus and/or both ovaries.
* any condition (including language barrier) that precludes patient's ability to comply with study requirements including completion of study.
* any condition that precludes the patient's ability or an assisting family member's ability to apply the medication drops or to sustain five minutes of pressure on the lacrimal ducts after drop application.
* concurrent enrollment in another clinical investigation medicinal product or device study is prohibited.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mines, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Ophthalmology Service at Walter Reed Army Medical Center, Washington DC from August 2007 to January 2011
Groups:
- Topical Avastin 1.0%: Each participant received topical Avastin to be applied to the affected eye either 2 or 4 times daily over a period of 3 weeks
Period: Overall Study
Arm/Group | Topical Avastin 1.0%
Started | 24
Completed | 20
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Topical Avastin 1.0%
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 52.3 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (Ocular and Systemic)
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Topical Avastin 1.0%
Number analyzed (Participants) | 20
participants | 0

2. Secondary Outcome: Size and Extent of Corneal Neovascularization
Description: computerized image analysis of the corneal photographs were used to measure the change in size and extent of corneal neovascularization from baseline.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Topical Avastin 1.0%
Number analyzed (Participants) | 20
percentage change | 27.9 (9.2)

ADVERSE EVENTS:
Groups:
- Topical Avastin 1.0%: Each participant received topical Avastin to be applied to the affected eye
Arm/Group | Topical Avastin 1.0%
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All materials that reflects the WRAMC affiliation must be approved and properly cleared before the material is submitted for public dissemination and publication. All publications whereby WRAMC is cited in the bylines will state on the cover page the following sample disclaimer: "The views expressed in this [article, book chapter, speech, presentation, etc.] are those of the author(s) and do not reflect the official policy of the Department of Army, Department of Defense, or U.S. Government."